CLINICAL TRIAL: NCT01277393
Title: Care of Critically Ill Patients Enteral Nutrition Guidelines for the Implementation of the Effectiveness of the Intervention
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Chin-Feng Huang, Nursing Department, Wanfang Hospital
Other Study IDs: 99058
Record Dates: First submitted 2011-01-12; First posted 2011-01-14 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: ICU Ill Patients; Enteral Nutrition Feeding
Keywords: Enteral nutrition feeding

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental Group
- Control Group

SUMMARY:
This study is to find out care of critically ill patients enteral nutrition guidelines for the implementation of the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients elder than 18 years of age
* (APACHE II) score > 15
* Patients expected to remain in ICU for more than 2 days

Exclusion Criteria:

* Patients that have consented to a Do-Not-Resuscitate document
* Patients not expected survive more than 2 days
* Patients that have returned to ICU due to their condition worsening after previously leaving ICU
* Patients that have transferred from ICU of other hospitals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ill patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Study Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Feng Huang, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan